CLINICAL TRIAL: NCT06242119
Title: Clinical Use of a J-PET Scanner Prototype Made of Plastic Scintilators
Brief Title: Clinical Application of the J-PET Scanner Prototype
Acronym: JPET2Clinic
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Collaborators: University Hospital in Krakow (Other)
Responsible Party: Principal Investigator, Ewa Stępień, PhD, Head of Department of Medical Physics, Institute of Physics, Jagiellonian University
Other Study IDs: MO 01.08.2023 J-PET
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Prostatic Hyperplasia; Prostatic Neoplasms; Prostate Cancer Metastatic; Neuroendocrine Tumors; Neuroendocrine Carcinoma
Keywords: positronium; PET; [18F]FDG; [18F]choline; [68Ga]Ga-DOTA-TATE; [68Ga]Ga-PSMA
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia; Neuroendocrine Tumors; Carcinoma, Neuroendocrine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- J-PET group: The patient is referred for a PET/CT scan, in accordance with recognized indications for examining the brain or the entire body.
  Interventions: Diagnostic Test: J-PET scan

INTERVENTIONS:
Diagnostic Test: J-PET scan — Diagnostic Test: Positron-Emission Tomography Imaging Examination of radiation distribution in the patient body after completing a routine examination on a PET diagnostic device. J-PET prototype tests will be carried out in patients who have undergone a classic PET examination after administration of [18F]FDG), [68Ga]Ga-PSMA, [18F]choline or [68Ga]Ga-DOTATATE). The duration of the additional exam will be approximately 20 minutes.

SUMMARY:
Positron emission tomography (PET), an advanced diagnostic imaging technique, exploits the annihilation of positrons (e+) to delineate pathological alterations within diseased tissues. Integral to PET scanners are detector systems that transform gamma photons into fluorescent photons, thereby gleaning insights into the energy, time, and spatial distribution of gamma photons emanating from positron-emitting radiopharmaceuticals. Conventional PET scanners, bear a significant financial burden primarily due to their reliance on LSO (lutetium oxyorthosilicate) or LYSO (lutetium yttrium oxyorthosilicate) scintillation crystals. The exorbitant cost and limited availability of these crystal scintillators impede the widespread adoption of PET scanners. In a departure from conventional PET technology, the prototype J-PET scanner employed in this trial employs plastic scintillators, characterized by unique physical properties. This prototype is further equipped with bespoke software enabling three-photon imaging based on the annihilation of ortho-positronium (o-Ps) generated within diseased tissue. This study delves into the clinical applicability of PET scanners employing plastic scintillators, particularly investigating the feasibility of PET imaging using plastic scintillators where gamma quanta interact by mechanisms other than the photoelectric effect. Furthermore, this study endeavors to contemporaneously acquire and analyze data related to the lifetime of ortho-positronium (o-P) atoms emanating from routine radiopharmaceuticals. Additionally, it seeks to validate the utilization of a novel diagnostic indicator, termed the &#34;positron biomarker,&#34; through a prospective study, comparing its efficacy to conventional diagnostic PET scanning methodologies.

DETAILED DESCRIPTION:
Positron emission tomography (PET) is currently one of the basic techniques enabling molecular imaging. This concept means imaging at the level of biochemical processes. The J-PET scanner is the world's first positron tomograph based on plastic strip scintillators to measure the lifetime of the ortho-positronium (o-Ps) atom. This is a modular scanner, designed and installed at the Department of Experimental Particle Physics and Applications of the Jagiellonian University in Krakow. The J-PET scanner is based on technology patented in 2014 and 2016.

Current PET cameras possess remarkable sensitivity, enabling the detection of changes in chemical concentration as subtle as 1E-11 moles. This unprecedented sensitivity allows for the visualization of metabolic alterations, neurotransmitter imbalances, or receptor system dysfunctions at an early stage, often before the onset of clinical symptoms in various diseases. The PET technique relies on radioisotopes that emit positrons, which are the antimatter counterparts of electrons. PET cameras, tasked with monitoring positron distribution, employ detector systems that capture the radiation generated during positron-electron annihilation. This annihilation process occurs in the emission of gamma ray photons, which are detected by the appropriate detector arrays. The computer system particularly records only those events that simultaneously trigger two detectors, ensuring high spatial resolution and precise anatomical localization of the annihilation events. Notably, positron annihilation may be preceded by the formation of positronium, a transient, quasi-stable bound state comprising an electron and its antiparticle, the positron. Due to the mutual arrangement of spins, two states of the positron are distinguished.

* When the electron and positron spins are parallel (triplet state ↑↑); this arrangement is called ortho-positronium (o-Ps). o-Ps decays (annihilation occurs) after an average vacuum lifetime of 142 nanoseconds [ns]. Annihilation produces three gamma ray photons.
* When the spins of the electron and positron are antiparallel (singlet state ↑↓) - the system is called para-positronium (p-Ps). Annihilation produces two gamma-ray photons with an average vacuum lifetime of 125 picoseconds [ps], or 1,136 times shorter.

Distinct from conventional PET scanners employed in diagnostic imaging, the J-PET scanner boasts three remarkable features:

1. Plastic Scintillation: unlike standard PET scanners that use expensive scintillation crystals, the J-PET scanner utilizes plastic scintillators, significantly lowering its cost and making it more affordable.
2. Modular Design: J-PET's modular design allows for easy customization to fit different patient sizes and can be expanded to a whole-body PET scanner. This flexibility caters to a wide range of patient populations and diagnostic needs.
3. Positronium Biomarker: J-PET expands the scope of PET imaging by introducing the detection and analysis of o-Ps.

Ad. 1. Conventional PET scanners use crystal detectors that detect gamma rays using the photoelectric effect. More expensive PET scanners use LSO, LYSO, or BGO crystals. New PET scanners use plastic detectors that detect gamma rays using Compton scattering. This allows for cheaper scanners with the same or better image quality.

Ad. 2. Thanks to the modular design and the use of strip scintillators, the time-of-flight (ToF) parameter is also used to improve image quality or obtain images of the same quality in a shorter examination because it reduces noise.

Ad.3. This capability opens up the possibility of utilizing a novel diagnostic biomarker that holds promising potential but remains underexplored in PET technology. Positronium imaging is applied only in the J-PET scanner. The PET technique uses radioisotopes that emit positron radiation (beta+). Traditional PET scanners image the distribution of gamma ray photons produced by the annihilation of an electron (e-) and a positron (e+). Annihilation may be preceded by the appearance of a positronium atom, which occurs in approximately 30-40% of all annihilations occurring in the patient body.

Working hypothesis:

The J-PET scanner is based on technology using plastic scintillators. If its clinical usefulness is proven, the development of this imaging method may significantly reduce the costs and increase the availability of PET/CT imaging.

Moreover, the J-PET tomograph allows us to determine a new diagnostic indicator, which is the lifetime of positronium atoms.

Aim of the study:

This study aims to demonstrate the clinical feasibility of PET scanners based on plastic scintillators, specifically investigating the performance of three-photon imaging and the use of positronium as a diagnostic biomarker. If the J-PET method allows to record the distribution of a chemical substance acting as a radiopharmaceutical with greater accuracy and - independently, it is possible to record the o-Ps lifetime depending on the biochemical composition of the environment, which is an additional parameter - not yet used in medical imaging.

ELIGIBILITY:
Inclusion Criteria:

* The patient is referred for a PET/CT scan, in accordance with recognized indications for examining the entire body.
* Age over 18 years
* Informed, voluntary consent to participate in the study

Exclusion Criteria:

* Pregnant women, breastfeeding women
* People with a previously diagnosed allergy to radiopharmaceuticals
* Age under 18 years
* Lack of cooperation with the patient
* Lack of informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group will include a maximum of 25 patients aged > 18 years referred for PET/CT examination using [68Ga]Ga-DOTA-TATE or [68Ga]Ga-PSMA or [18F]FDG or [18F ]choline in accordance with recognized oncological clinical indications to the Department of Nuclear Medicine, O/K Department of Endocrinology, Oncological Endocrinology and Nuclear Medicine of the University Hospital in Krakow, who give informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Intraclass correlation coefficient (ICC) | Initial analyzes will last 12 weeks
  ICC for Cancer Stage using the union for international cancer control (UICC) TNM (T= tumor, N= nodal stage, M = metastasis) System (8th Edition) for plastic scanner positron emission and computed tomography (J-PET/CT) exams compared to the standard of care (SOC) full-dose PET/CT as assessed by a panel of physicians

SECONDARY OUTCOMES:
Image quality | after 3 months following scan
  Composite outcome assessing image quality in terms of tumour to background ratio (TBR) and signal to noise (SNR), defined as the reciprocal coefficient of variation (COV) for J-PET/CT compared to the standard of care PET/CT
Subjective quality | after 3 months following scan
  Image quality (subjective) as rated by five independent nuclear medicine physicians on a five-point Likert scale (1= unacceptable, 2=poor, 3=moderate, 4=good, 5=high) for J-PET/CT compared to the standard of care PET/CT
Agreement | after 3 months following scan
  Inter-reader agreement for the primary outcome (UICC cancer stage) shall be compared between J-PET/CT and the standard of care PET/CT
Diagnostic accuracy | after 6 months following scan
  Assessment of the positive predictive value (PPV) for J-PET/CT compared to the standard of care PET/CT for patients who undergo surgery or biopsy and where histopathological confirmation of true positive (TP) and false positive (FP) findings are available

CONTACTS AND LOCATIONS:
Overall Officials: Marta Opalinska, MD, PhD, Principal Investigator — Department of Endocrinology and Nuclear Medicine, University Hospital in Krakow; Pawel Moskal, PhD, Study Chair — Jagiellonian University; Ewa Stepien, PhD, Study Director — Jagiellonian University
Locations (1):
- Department of Endocrinology and Nuclear Medicine, University Hospital in Krakow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moskal P, Dulski K, Chug N, Curceanu C, Czerwinski E, Dadgar M, Gajewski J, Gajos A, Grudzien G, Hiesmayr BC, Kacprzak K, Kaplon L, Karimi H, Klimaszewski K, Korcyl G, Kowalski P, Kozik T, Krawczyk N, Krzemien W, Kubicz E, Malczak P, Niedzwiecki S, Pawlik-Niedzwiecka M, Pedziwiatr M, Raczynski L, Raj J, Rucinski A, Sharma S, Shivani, Shopa RY, Silarski M, Skurzok M, Stepien EL, Szczepanek M, Tayefi F, Wislicki W. Positronium imaging with the novel multiphoton PET scanner. Sci Adv. 2021 Oct 15;7(42):eabh4394. doi: 10.1126/sciadv.abh4394. Epub 2021 Oct 13. PMID 34644101
- [Background] Moskal P, Stepien EL. Prospects and Clinical Perspectives of Total-Body PET Imaging Using Plastic Scintillators. PET Clin. 2020 Oct;15(4):439-452. doi: 10.1016/j.cpet.2020.06.009. Epub 2020 Jul 29. PMID 32739047
- [Background] Moskal P, Kubicz E, Grudzien G, Czerwinski E, Dulski K, Leszczynski B, Niedzwiecki S, Stepien EL. Developing a novel positronium biomarker for cardiac myxoma imaging. EJNMMI Phys. 2023 Mar 24;10(1):22. doi: 10.1186/s40658-023-00543-w. PMID 36959477
- [Background] Dadgar M, Parzych S, Baran J, Chug N, Curceanu C, Czerwinski E, Dulski K, Elyan K, Gajos A, Hiesmayr BC, Kaplon L, Klimaszewski K, Konieczka P, Korcyl G, Kozik T, Krzemien W, Kumar D, Niedzwiecki S, Panek D, Perez Del Rio E, Raczynski L, Sharma S, Shivani S, Shopa RY, Skurzok M, Stepien EL, Tayefi Ardebili F, Tayefi Ardebili K, Vandenberghe S, Wislicki W, Moskal P. Comparative studies of the sensitivities of sparse and full geometries of Total-Body PET scanners built from crystals and plastic scintillators. EJNMMI Phys. 2023 Oct 11;10(1):62. doi: 10.1186/s40658-023-00572-5. PMID 37819578
- [Background] Moskal P, Kisielewska D, Curceanu C, Czerwinski E, Dulski K, Gajos A, Gorgol M, Hiesmayr B, Jasinska B, Kacprzak K, Kaplon L, Korcyl G, Kowalski P, Krzemien W, Kozik T, Kubicz E, Mohammed M, Niedzwiecki S, Palka M, Pawlik-Niedzwiecka M, Raczynski L, Raj J, Sharma S, Shivani, Shopa RY, Silarski M, Skurzok M, Stepien E, Wislicki W, Zgardzinska B. Feasibility study of the positronium imaging with the J-PET tomograph. Phys Med Biol. 2019 Mar 7;64(5):055017. doi: 10.1088/1361-6560/aafe20. PMID 30641509
- [Background] Huang B, Li T, Arino-Estrada G, Dulski K, Shopa RY, Moskal P, Stepien E, Qi J. SPLIT: Statistical Positronium Lifetime Image Reconstruction via Time-Thresholding. IEEE Trans Med Imaging. 2024 Jun;43(6):2148-2158. doi: 10.1109/TMI.2024.3357659. Epub 2024 Jun 3. PMID 38261489
- See also: Description Patent US8859973B2: Strip device and method for determining the location and time of reaction of the gamma quanta and the use of the device to determine the location and time of reaction of the gamma quanta in positron emission tomography — https://patents.google.com/patent/US8859973B2/en?oq=US+8%2c859%2c973
- See also: P. Moskal, "Positronium Imaging," 2019 IEEE Nuclear Science Symposium and Medical Imaging Conference (NSS/MIC), Manchester, UK, 2019, pp. 1-3 — https://ieeexplore.ieee.org/document/9059856
- See also: Description Patent US9804274B2:Hybrid TOF-PET/CT tomograph comprising polymer strips made of scintillator material — https://patents.google.com/patent/US9804274B2/en?q=(positronium)&inventor=moskal&oq=moskal+positronium